CLINICAL TRIAL: NCT03060772
Title: A Study of Pleiotropic Pioglitazone Effects on the Alcoholic Lung (APPEAL Study)
Acronym: APPEAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was suspended in 2020 due to COVID-19 pandemic as a result of recruitment challenges and the inability to conduct all study procedures (e.g., bronchoscopy) per protocol. In late 2021 the decision was made to not re-open the study.
Sponsor: Emory University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, David M. Guidot, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00071908; 1R01AA025857 (NIH)
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Alcoholism
Keywords: Pulmonary Medicine; Oxidative Stress; Pioglitazone; Immunology; Addictive/Compulsive Behavior
MeSH Terms: conditions — Alcoholism; Compulsive Behavior | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: Individuals with alcohol use disorder will be randomized to receive the study medication, pioglitazone, or no medication (12 in each group). A third group of healthy individuals who do not have an alcohol use disorder will also be enrolled to serve as an additional comparison group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Alcohol use disorder - Pioglitazone Treatment (Experimental): Participants with alcohol use disorder randomized to this group will receive pioglitazone. Study procedures include a bronchoscopy at baseline and an additional bronchoscopy after taking the study medication for 2 to 4 weeks.
  Interventions: Drug: Pioglitazone
- Alcohol use disorder - No Pioglitazone (No Intervention): Participants with alcohol use disorder randomized to this group will receive their usual care but will not receive pioglitazone. Study procedures include a bronchoscopy at baseline and an additional bronchoscopy 2 to 4 weeks later.
- Healthy controls without alcohol use disorder (No Intervention): Healthy individuals who do not have alcohol use disorder will be enrolled will serve as a control group. Healthy controls will be a matched to participants receiving the treatment based on age, gender, and smoking status. This group will have a single bronchoscopy.

INTERVENTIONS:
Drug: Pioglitazone — Participants will take 30 mg of pioglitazone once daily for a total of two to four weeks for those randomized to therapy, until the next bronchoscopy is performed. Participants will receive 14 to 28 tablets of active pioglitazone, which is enough to complete the minimum 14-day course of therapy.
  Other Names: Actos
  Arms: Alcohol use disorder - Pioglitazone Treatment

SUMMARY:
This study is a single center, open-label, randomized clinical trial to determine the effect of pioglitazone (PIO) treatment on alveolar macrophage immune function, redox stress, and NADPH oxidase expression in outpatient alcoholic subjects. The researchers will recruit a cohort of otherwise healthy patients with an alcoholic use disorder from the Substance Abuse Treatment Program at the Atlanta Veterans Affairs (VA) Medical Center and randomize them to receive the usual treatment for two to four weeks or to the usual treatment plus PIO treatment for two to four weeks. There will also be a healthy control group (matched on age, gender, and smoking status) that will receive no treatment. To measure the effect of pioglitazone, participants will undergo a bronchoscopy before taking the study drug and then again 2-4 weeks later to look for changes. The bronchoscopy will allow researchers to obtain fluid from the lungs to see how well their immune cells respond to bacteria by determining phagocytic capacity.

DETAILED DESCRIPTION:
Alcohol abuse is a major burden on society and an enormous problem in the veteran population. Many people are aware that chronic alcohol ingestion can cause serious health problems like liver injury and brain damage but chronic alcohol consumption can also hurt the lungs. People who regularly drink more than the daily maximum levels recommended by the Centers for Disease Control and Prevention (CDC) (1 drink per day for women or 2 drinks per day for men) are more likely to suffer from pneumonia and acute lung injuries.

The primary goal of this clinical research study is to determine if a Food and Drug Administration (FDA) approved diabetes drug, called pioglitazone, can improve the lung immune defenses in otherwise healthy alcoholics. There is strong evidence from experimental animal models that pioglitazone preserves lung health even during daily alcohol ingestion.

This National Institutes of Health (NIH) funded project will recruit veterans who are patients at the Atlanta VA Hospital. Half of the participants will be randomly assigned to receive pioglitazone and half will be assigned to receive no treatment. Participants assigned to pioglitazone will take the pill once per day for two to four weeks. To measure the effect of pioglitazone, participants will undergo a procedure called a bronchoscopy before taking the study drug and then again 2-4 weeks later to look for changes. The bronchoscopy will allow researchers to obtain fluid from the lungs to see how well their immune cells respond to bacteria (by determining phagocytic capacity). The researchers also plan to enroll 12 healthy veteran patients who do not drink. These participants will undergo a one-time bronchoscopy and no other visits will be required of them.

The findings from this study will guide future, larger scale clinical trials to determine if pioglitazone can be used in the clinical setting to improve outcomes in alcoholics who develop pneumonia or acute lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Active alcohol use disorder, with last alcoholic drink within 8 days of randomization (for those in the alcohol use disorder arms)

Exclusion Criteria:

* History of diabetes
* History of heart failure
* History of cirrhosis of the liver
* Elevation of liver enzymes greater than 2.5 times upper limit of normal
* History of bladder cancer
* Primary substance of abuse is something other than alcohol
* Current abnormal chest x-ray or other evidence of significant lung disease
* HIV-positive
* Renal impairment, defined as glomerular filtration rate (GFR) <60
* Current pregnancy or planning to become pregnant in the next 6 months
* Currently on pioglitazone treatment for another reason
* Contraindication to treatment with pioglitazone
* Any active and uncontrolled medical problem that may negatively impact the study results
* Currently on an oral steroid or inhaled corticosteroid
* History of profound psychiatric problems, poor compliance, or other psycho-social issues that may negatively impact participation
* Inability to give informed consent (i.e., limited cognitive capacity)
* Non-English speaking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Change in phagocytic index | Baseline, After 2-4 weeks
  The change in phagocytic index will be determined between the alcohol use disorder study arms to examine the effect of PIO treatment. Phagocytic index of the alveolar macrophage is the rate at which particles are cleared from a culture. The phagocytic index is a well-established marker of immune function and its improvement with pioglitazone (PIO) treatment would indicate reversal of the alcoholic lung phenotype. The phagocytic index will be measured in bronchoalveolar lavage (BAL) fluids.

SECONDARY OUTCOMES:
Change in nicotinamide adenine dinucleotide phosphate-oxidase (NADPH oxidase) | Baseline, After 2-4 weeks
  The change in nicotinamide adenine dinucleotide phosphate-oxidase (NADPH oxidase) will be determined between the alcohol use disorder study arms to examine the effect of PIO treatment. Nicotinamide adenine dinucleotide phosphate-oxidase (NADPH oxidase) is an enzyme complex. NADPH oxidases are the primary sources of oxidative stress in the alveolar macrophage. Chronic alcohol consumption causes pulmonary oxidative stress via increased expression and activity of NADPH oxidases. NADPH oxidases will be measured in bronchoalveolar lavage (BAL) fluids.
Change in alveolar macrophage oxidative stress | Baseline, After 2-4 weeks
  The change in alveolar macrophage oxidative stress will be determined between the alcohol use disorder study arms to examine the effect of PIO treatment. The alveolar macrophage plays a crucial role in lung immunity by protecting the individual from developing respiratory infections such as pneumonia. Alcohol-induced oxidative stress impairs the ability of the alveolar macrophage to function normally. A decrease in alveolar oxidative stress with pioglitazone treatment would indicate that the treatment is having a positive impact. This outcome will be measured in bronchoalveolar lavage (BAL) fluids.
Change in redox couple glutathione/glutathione disulfide (GSH/GSSG) | Baseline, After 2-4 weeks
  The change in redox couple glutathione/glutathione disulfide (GSH/GSSG) will be determined between the alcohol use disorder study arms to examine the effect of PIO treatment. Glutathione (GSH)/glutathione disulfide (GSSG) is a redox (a chemical reaction) which is frequently measured as an indicator of oxidative stress. The antioxidant GSH reduces to GSSG and in a healthy state there is greater than 90% GSH to less than 10% GSSG. Chronic alcohol consumption causes pulmonary oxidative stress via decreased levels of GSH. GSH and GSSG will be measured in bronchoalveolar lavage (BAL) and exhaled breath condensate (EBC) fluids.
Change in cysteine/cystine (Cys/CySS) redox potential | Baseline, After 2-4 weeks
  The change in cysteine/cystine (Cys/CySS) redox potential will be determined between the alcohol use disorder study arms to examine the effect of PIO treatment. Cysteine (Cys)/cystine (CySS) is a redox (a chemical reaction) regulating a variety of biological processes. CySS is the oxidized form of Cys and the ratio is sensitive to alcohol abuse, among other environmental exposures. Cys and CySS will be measured in bronchoalveolar lavage (BAL) and exhaled breath condensate (EBC) fluids.
Comparison of nicotinamide adenine dinucleotide phosphate-oxidase (NADPH oxidase) | Baseline (control group), After 2-4 weeks (treatment group)
  Nicotinamide adenine dinucleotide phosphate-oxidase (NADPH oxidase) will be compared between the PIO treatment arm and the healthy control arm to determine if PIO treatment leads to normal function. Nicotinamide adenine dinucleotide phosphate-oxidase (NADPH oxidase) is an enzyme complex. NADPH oxidases are the primary sources of oxidative stress in the alveolar macrophage. Chronic alcohol consumption causes pulmonary oxidative stress via increased expression and activity of NADPH oxidases. NADPH oxidases will be measured in bronchoalveolar lavage (BAL) fluids.
Comparison of alveolar macrophage oxidative stress | Baseline (control group), After 2-4 weeks (treatment group)
  Alveolar macrophage oxidative stress will be compared between the PIO treatment arm and the healthy control arm to determine if PIO treatment leads to normal function. The alveolar macrophage plays a crucial role in lung immunity by protecting the individual from developing respiratory infections such as pneumonia. Alcohol-induced oxidative stress impairs the ability of the alveolar macrophage to function normally. A decrease in alveolar oxidative stress with pioglitazone treatment would indicate that the treatment is having a positive impact. This outcome will be measured in bronchoalveolar lavage (BAL) fluids.
Comparison of redox couple glutathione/glutathione disulfide (GSH/GSSG) | Baseline (control group), After 2-4 weeks (treatment group)
  Redox couple glutathione/glutathione disulfide (GSH/GSSG) will be compared between the PIO treatment arm and the healthy control arm to determine if PIO treatment leads to normal function. Glutathione (GSH)/glutathione disulfide (GSSG) is a redox (a chemical reaction) which is frequently measured as an indicator of oxidative stress. The antioxidant GSH reduces to GSSG and in a healthy state there is greater than 90% GSH to less than 10% GSSG. Chronic alcohol consumption causes pulmonary oxidative stress via decreased levels of GSH. GSH and GSSG will be measured in bronchoalveolar lavage (BAL) and exhaled breath condensate (EBC) fluids.
Comparison of cysteine/cystine (Cys/CySS) redox potential | Baseline (control group), After 2-4 weeks (treatment group)
  Cysteine/cystine (Cys/CySS) redox potential will be compared between the PIO treatment arm and the healthy control arm to determine if PIO treatment leads to normal function. Cysteine (Cys)/cystine (CySS) is a redox (a chemical reaction) regulating a variety of biological processes. CySS is the oxidized form of Cys and the ratio is sensitive to alcohol abuse, among other environmental exposures. Cys and CySS will be measured in bronchoalveolar lavage (BAL) and exhaled breath condensate (EBC) fluids.

CONTACTS AND LOCATIONS:
Overall Officials: David Guidot, MD, Principal Investigator — Emory University
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT03060772/ICF_000.pdf